CLINICAL TRIAL: NCT07024472
Title: NIBP Cuff Material Comparison Study
Brief Title: NIBP Cuff Comparison Study
Status: Completed | Type: Observational
Sponsor: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 11897689627
Record Dates: First submitted 2025-03-31; First posted 2025-06-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-03

CONDITIONS: Blood Pressure; Blood Pressure Measurement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of the study is to compare NIBP cuff materials and their effect on the measurement results.

DETAILED DESCRIPTION:
Non-invasive blood pressure measurement is based on the estimation of blood pressure by using cuffs. Because the accuracy in blood pressure measurement is essential to monitor patients, the reliability of non-invasive sphygmomanometers is required by internationally recognized standards. New NIBP standard ISO 81060-2 AMD2 highlights the impact of cuff materials and construction on NIBP clinical accuracy. This study is designed to gather evidence that different cuffs provide equally comparable NIBP measurement results

ELIGIBILITY:
Inclusion Criteria:

1. Age >= 18 years to 65 years
2. Are able and willing to comply with the study procedures.
3. Are able and willing to provide written informed consent to participate.
4. A cuff of same size is applicable to both arms (difference between the limbs should be less than 2cm)
5. Blood pressure needs to be measurable from both arms.

Exclusion Criteria:

1. Are pregnant.
2. Are breastfeeding.
3. Have participated in the study. No subject may participate more than once.
4. Have an AV fistula.
5. Have acute infection.
6. Have subject reported arrythmias.
7. PI or designee decision due to subject health conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-06-23 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | From admission to discharge
  The primary outcome is to collect NIBP measurement data from subjects in laboratory setting to show equivalency of the different NIBP Cuff.

CONTACTS AND LOCATIONS:
Locations (1):
- Metropolia University of Applied Sciencies, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No